CLINICAL TRIAL: NCT04283448
Title: Gut Microbiota Dependent and Independent Impacts of Dietary Pulses on Pre- and Postprandial Metabolism and Inflammation in Overweight/Obese Humans
Brief Title: Impacts of Lentils on Metabolism and Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montana State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 58-3060-9-040
Record Dates: First submitted 2020-02-05; First posted 2020-02-25 (Actual); Results first posted 2024-12-13 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Hypertriglyceridemia; Inflammation; Waist, Hypertriglyceridemic
MeSH Terms: conditions — Hypertriglyceridemia; Inflammation; Hypertriglyceridemic Waist

STUDY DESIGN:
Intervention Model Description: This study will utilize a parallel intervention of meals with 0.66 cups of lentils each day versus macronutrient-matched (not including fiber) meals with 0 cups of lentils each day for 12 weeks in OW/OB adults with demonstrated risk for T2D and CVD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lentil (Experimental): 0.66 cups lentils
  Interventions: Behavioral: Dietary Lentil
- Control (Sham Comparator): 0.0 cups lentils
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Dietary Lentil — Participants in the Lentil arm of the study will consume midday meals containing 0.66 cups of lentils seven days per week for 12 weeks.
  Arms: Lentil
Behavioral: Control — Participants in the Control arm of the study will consume midday meals containing 0.00 cups of lentils seven days per week for 12 weeks.
  Arms: Control

SUMMARY:
The overall goal of this investigation is to determine gut microbiome dependent and independent impacts of pulse consumption on metabolic resilience and metabolic risk profiles for type 2 diabetes (T2D) and cardiovascular disease (CVD) risk. Specifically, pulse crop consumption has unrealized potential to fundamentally alter how the body responds to disease promoting metabolic stresses of postprandial triglyceride and inflammation responses. The specific objectives are to (1) Determine the impact of green lentil consumption on postprandial triglyceride (TG) and inflammation responses to a high-fat meal challenge. (2) Determine the extent to which the gut microbiome and changes in the gut microbiome induced by pulse consumption influence health impacts (3) Measure metabolomic profiles to elucidate underlying mechanisms linking pulse consumption to improved health. To achieve these objectives investigators will determine the effects of green lentil on high impact risk factors of large postprandial triglyceride excursions and inflammation, composition of and changes in the gut microbiomes, and both gut and serum metabolomes in overweight/obese (OW/OB) individuals with elevated risk. The 12-week intervention will consist of consumption of 4.6 or 0 cups of pulses per week across 7 pre-made meals (matched for macronutrient content (except fiber) provided to experimental and control groups. The following hypotheses will be tested in the proposed investigation:

H1: Lentil consumption lower postprandial TG and inflammation responses and improve overall metabolic health.

H2: Characteristics of the gut microbiome and changes in the gut microbiome induced by lentil consumption substantially influence health impacts of pulse consumption.

H3: Features of the fecal and serum metabolomes distinguishing lentil and control treatments correspond to metabolic pathways elucidating potential gut microbiome dependent and independent mechanisms linking pulse consumption to improved health.

DETAILED DESCRIPTION:
Investigators will utilize a parallel intervention of lentil versus macronutrient-matched (not including fiber) control treatment for 12 weeks in OW/OB adults with demonstrated risk for T2D and CVD. Experimental diets will be provided to participants in the form of pre-made midday meals to exploit the second meal effect and lower caloric intake at the evening meal. Pre- and post-intervention assessments will be made for the following variables: makeup of the gut microbiome (microbial species and relative abundance), gut metabolome, postprandial response of TG, inflammatory cytokines, and serum metabolome to a high-fat meal challenge (established inflammation stimulus), fasting serum glucose, lipid, insulin, inflammation markers and metabolome, blood pressure, and anthropometric measures including weight, body composition, waist circumference, and quantity of visceral adipose tissue. Habitual diet will be measured so that these variables can be used to aid in our characterization of participants and aid in analysis and interpretation of data.

Procedures:

Postprandial lipidemic and inflammation responses: High-fat meal challenges with 40 to 100 g of dietary fat are an established laboratory test to measure both postprandial triglyceridemic and inflammation responses. Investigators have used a 50 g dose of fat delivered in the form of butter on toast on > 50 individuals because this particular dose is effective at discriminating between low versus high TG and inflammation responders. In brief, participants will report to the laboratory after an overnight fast, an indwelling venous catheter will be placed in an antecubital vein, and blood samples will be collected before, and 1, 2, 3, 4, and 5 hours following ingestion of the high-fat meal. Samples will be analyzed in real time for TG (and full lipid panel plus glucose) using a clinical chemistry analyzer (Piccolo xpress), while serum samples will be aliquoted and stored at -80 C until analysis for inflammatory cytokines, metabolomics, and insulin. Investigators will measure inflammatory cytokines (TNF-α, IFN-y, interleukin (IL)-1β, IL-6 IL-17, IL-23, IL-10, and granulocyte macrophage colony stimulating factor (GM-CSF)) using high-sensitivity Luminex multiplexing technology (Bio-Rad Bio-Plex® 200 HTS) prepared by Millipore.

Dietary intervention: Using methods established for an ongoing CRT with lentils, investigators will prepare 7 meals per participant per week to deliver a dose of 4.6 or 0 cups of lentils per week for the experimental and control groups. Meals are matched for macronutrient content (except for fiber), and ground turkey or chicken replaces lentils in the control meals. Dietary intervention will be 12 weeks in length with a possible extension to 13 weeks if participants either 1) miss 3 or more meals in a row at any point during the intervention or 2) miss any meals at all in the last week of the intervention prior to their final visit. To keep the meal intervention period between 12 and 13 weeks, participants will be dropped from the study if meal adherence failures result in more than a one week intervention extension.

Participants will be instructed to consume food provided for their midday meal, and then to proactively reduce portion sizes and to not eat beyond fullness at the evening meal. This strategy exploits the satiety effect of pulses at the midday meal and the 'second meal effect' in which volitional consumption is reduced at the next meal, the evening meal. Each participant will be surveyed once weekly to determine whether they consumed the experimental meal that day, their perceptions of hunger, fullness, satiety, and satisfaction with that day's meal (at 4:00 pm), and their gastrointestinal comfort (level of bloating, flatulence, cramping, and comfort) throughout the day (at 8:00 pm). This methodology has been successfully implemented in our ongoing study to demonstrate that lentil meals are equally pleasing, produce greater satiety, and are well-tolerated.

Gut microbiome analysis: Bulk DNA will be extracted from fecal samples using the Powersoil® DNA Isolation Kit (Mo Bio Laboratories Inc.). DNA will be shipped overnight to the University of Michigan, Center for Microbial Systems, for Illumina MiSeq amplicon sequencing of the 16S V4 variable region. Raw sequencing reads will be processed and curated using the mothur (v.1.39.5) software package, following the mothur MiSeq standard operating procedure, potentially chimeric sequences will be identified and removed using the Uchime (v4.2.40) algorithm, and taxonomic classifications will be assigned using the Bayesian classifier of the Ribosomal Database Project, and operational taxonomic units (OTUs) will be assigned in mothur using the VSEARCH distance-based clustering algorithm at the 97% sequence similarity threshold.

Metabolomic analysis: Samples will be analyzed by high resolution liquid chromatography mass spectrometry (LCMS). Hydrophilic interaction chromatography (HILIC) and reverse-phase (RP) columns will be used for deep coverage. Metabolite identification will use fragmentation pattern matching, authentic standards and database matching with METLIN and the Human Metabome Database (HDB). Novel features of significant interest will be characterized with liquid chromatography mass spectrometry solid phase extraction nuclear magnetic resonance (LCMS-SPE-NMR). Pathway analysis will use XCMS and mummichog.

Dietary analysis. Long-term dietary habits may create adaptations that influence the response to the short-term supplementation of Aronia and lentil. This study will use the most recent version (2018) of the web-based Diet History Questionnaire (DHQ III), a food frequency questionnaire designed for adults 19 and older, developed by staff at the Risk Factor Monitoring and Methods Branch (RFMMB) of the NIH National Cancer Institute. The outputs of the DHQ III include carbohydrate constituents, carotenoids and tocopherols, dietary constituents from supplements, fats, fatty acids and cholesterol, macronutrients and energy, minerals, protein constituents, and vitamins are dietary constituents and food groups available in the DHQ III output files.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference > 35 inches for women and > 40 inches for men
* Non-fasting serum triglyceride concentration > 175 mg/dl

Exclusion Criteria:

* Allergy to wheat
* Taking medication that will influence cholesterol, lipids, or inflammation
* Pregnant or use of hormonal contraceptive method
* Have diabetes, a pacemaker, or other health conditions that may interfere with the study outcomes
* Planning to undergo a weight loss intervention or change in exercise regimen

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2023-11-19 (Actual); Study Completion 2023-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Miles, PhD, Principal Investigator — Montana State University
Locations (1):
- Nutrition Research Laboratory, Bozeman, Montana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lentil | Control
Started | 20 | 18
Completed | 20 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lentil | Control | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.65 (11.52) | 43.20 (14.01) | 47.11 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 35
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 18 | 17 | 35
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 17 | 36
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change in Postprandial Serum Triglyceride
Description: Area under the curve for serum triglyceride concentration calculated from 0 - 5 hours post consumption of a meal containing 50 g of fat. Value reported as the change from baseline to 12 weeks post intervention (Value at 12 weeks minus value at baseline).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmol*hr/L
Arm/Group | Lentil | Control
Number analyzed (Participants) | 20 | 18
mmol*hr/L | -0.1 (1.5) | 0.2 (1.8)

2. Primary Outcome: Change in Postprandial Serum Glucose
Description: Area under the curve for serum glucose concentration calculated from 0 - 5 hours post consumption of a meal containing 50 g of fat. Value reported as the change from baseline to 12 weeks post intervention (Value at 12 weeks minus value at baseline)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmol*hr/L
Arm/Group | Lentil | Control
Number analyzed (Participants) | 20 | 18
mmol*hr/L | -0.7 (1.4) | 0.1 (1.8)

3. Primary Outcome: Change in Postprandial Serum Inflammatory Cytokines
Description: Area under the curve for inflammatory cytokine (tumor necrosis factor-alpha, interleukin-(IL)1beta, IL-6, IL-10, IL-17, IL-23, interferon-gamma, and granulocyte macrophage-colony stimulating factor) concentration calculated from 0 - 5 hours post consumption of a meal containing 50 g of fat. Value reported as the change in AUC for each cytokine from baseline to 12 weeks post intervention (Value at 12 weeks minus value at baseline).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: pg*hr/ml
Arm/Group | Lentil | Control
Number analyzed (Participants) | 20 | 18
pg*hr/ml
  tumor necrosis factor-alpha | -7.59 (21.85) | 3.07 (9.37)
  IL-1beta | -4.06 (9.94) | 1.09 (3.92)
  IL-6 | -12.42 (31.92) | 0.09 (3.93)
  IL-10 | -43.64 (133.11) | 8.69 (38.50)
  IL-17 | -27.07 (83.07) | 13.82 (31.64)
  IL-23 | -234.36 (941.87) | 122.67 (731.23)
  interferon-gamma | -27.20 (438.32) | 6.99 (434.06)
  granulocyte macrophage-colony stimulating factor | -24.35 (67.97) | -77.16 (482.39)

4. Primary Outcome: Change in Fasting Serum Lipids and Glucose
Description: Concentration of HDL, LDL, TG, and glucose in the serum after an overnight fast. Value reported as the change in value from baseline to 12 weeks post intervention (Value at 12 weeks minus value at baseline).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Lentil | Control
Number analyzed (Participants) | 20 | 18
mmol/L
  Cholesterol | -0.11 (0.50) | 0.36 (0.43)
  HDL | -0.07 (0.15) | 0.10 (0.14)
  LDL | -0.03 (0.43) | 0.30 (0.36)
  Triglyceride | -0.06 (0.73) | -0.21 (0.54)
  Glucose | -0.06 (0.34) | -0.05 (0.44)

5. Primary Outcome: Change in Fasting Inflammatory Cytokines
Description: Concentration of inflammatory cytokines (tumor necrosis factor-alpha, interleukin-(IL)1beta, IL-6, IL-10, IL-17, IL-23, interferon-gamma, and granulocyte macrophage-colony stimulating factor) in the serum after an overnight fast. Value reported as the change from baseline to 12 weeks post intervention (Value at 12 weeks minus value at baseline)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Lentil | Control
Number analyzed (Participants) | 20 | 18
pg/ml
  tumor necrosis factor-alpha | 1.47 (4.17) | -0.76 (1.88)
  IL-1beta | 0.65 (2.05) | 0.04 (0.78)
  IL-6 | 2.20 (5.52) | 0.26 (1.79)
  IL-10 | 3.46 (12.93) | 0.62 (12.72)
  IL-17 | 3.56 (12.62) | -0.84 (4.93)
  IL-23 | -28.54 (527.21) | -12.27 (129.2)
  interferon-gamma | 9.69 (143.72) | 11.67 (85.84)
  granulocyte macrophage-colony stimulating factor | 3.00 (24.99) | -4.53 (17.42)

6. Secondary Outcome: Change in Body Fat Composition
Description: Change in % Body Fat from baseline to 12 weeks post intervention (Value at 12 weeks minus value at baseline)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of Body Fat
Arm/Group | Lentil | Control
Number analyzed (Participants) | 20 | 18
percentage of Body Fat | -1.2 (6.4) | 0.55 (1.9)

7. Secondary Outcome: Change in Visceral Adipose Tissue
Description: Change in the quantity of adipose tissue located within the abdominal compartment from baseline to 12 weeks post intervention (Value at 12 weeks minus value at baseline)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Lentil | Control
Number analyzed (Participants) | 20 | 18
Liters | 0.08 (0.92) | 0.17 (0.63)

8. Secondary Outcome: Change in Body Mass Index (BMI)
Description: Change in BMI (kg/m^2) from baseline to 12 weeks post intervention (Value at 12 weeks minus value at baseline).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: kg of mass per meter of height squared
Arm/Group | Lentil | Control
Number analyzed (Participants) | 20 | 18
kg of mass per meter of height squared | -0.43 (1.21) | -0.02 (0.96)

9. Secondary Outcome: Perceptions of Hunger, Fullness, Satiety, and Satisfaction After Mid-day Meal During the Intervention
Description: Ratings of hunger, fullness, satiety, satisfaction, desire to eat, and desire to consume additional food in response to mid-day meal consumption during the 12-week intervention. Ratings were scored on a scale of 0 to 10 with 0 representing no feelings of hunger, fullness, satiety, satisfaction, desire to eat, or consume additional food and 10 representing maximal feelings of hunger, fullness, satiety, satisfaction, desire to eat, or consume additional food. Reported values represent the average from all survey responses collected over the duration of the 12-week intervention period.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale (0=lowest, 10=highest)
Arm/Group | Lentil | Control
Number analyzed (Participants) | 20 | 18
units on a scale (0=lowest, 10=highest)
  Hunger (lower scores indicate low hunger after consuming meal) | 3.6 (2.0) | 3.9 (2.1)
  Fullness (lower scores indicate low fullness after consuming meal) | 6.3 (2.3) | 6.2 (2.0)
  Satisfaction (lower scores indicate low satiety after consuming the meal) | 6.2 (2.1) | 6.1 (1.9)
  Desire to eat (lower scores indicate little desire to eat more food after consuming the meal) | 4.0 (2.2) | 4.2 (2.2)
  Amount of food that could be eaten (lower scores indicate that little food is desired) | 3.6 (1.9) | 4.0 (2.0)

10. Secondary Outcome: Gastrointestinal Symptoms of Bloating, Cramping, Discomfort, and Flatulence During the Intervention
Description: Ratings of the gastrointestinal symptoms of bloating, cramping, discomfort, and flatulence over the 12-week intervention. All symptoms were qualitatively ranked as "none", "mild", "moderate", or "severe" by participants. Numerical values were then assigned to all measures using a 4-point scale: (0 = none, 1 = mild, 2 = moderate, 3 = severe). Values reported represent the average from all surveys collected during the 12 week intervention.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lentil | Control
Number analyzed (Participants) | 20 | 18
score on a scale
  Flatulence (lower scores indicate less flatulence) | 0.9 (0.7) | 0.8 (0.9)
  Bloating (lower scores indicate less bloating) | 0.6 (0.8) | 0.7 (0.9)
  Cramping (lower scores indicate less cramping) | 0.2 (0.5) | 0.3 (0.7)
  Discomfort (lower scores indicate less abdominal discomfort) | 0.3 (0.6) | 0.4 (0.8)

11. Other Pre Specified Outcome: Change in Habitual Diet
Description: Healthy Eating Index (HEI) scores were obtained through DHQ III survey data output from before and after the 12 week intervention. Each category is scored on a scale of 0-5 or 0-10. For components of adequacy, high scores indicate higher intake of each component and are therefore desirable. For components of moderation, high scores indicate lower intake of each component and are therefore desirable. Total possible scores for components of adequacy are as follows: Total Fruits (5), Whole Fruits (5), Total Vegetables (5), Greens and Beans (5), Whole Grains (10), Dairy (10), Total Protein Foods (5), Seafood and Plant Proteins (5), Fatty acids (10). Total possible scores for components of moderation are as follows: Refined Grains (10), Sodium (10), Added sugar (10). Total HEI score is also reported as the sum of all components with a total possible score of 100 indicating healthiest possible diet. All values reported as the change in value from baseline to 12 weeks post intervention.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: HEI Scores from DHQIII
Groups:
- Control: 0 cups lentils
Arm/Group | Lentil | Control
Number analyzed (Participants) | 20 | 18
HEI Scores from DHQIII
  Total Fruits (0-5 score possible, higher indicating healthier score) | -0.1 (1.6) | -0.8 (1.5)
  Whole Fruits (0-5 score possible, higher indicating healthier score) | -0.1 (1.6) | -0.5 (1.3)
  Total Vegetables (0-5 score possible, higher indicating healthier score) | 0.6 (1.1) | 0.1 (1.1)
  Green and Beans (0-5 score possible, higher indicating healthier score) | 0.8 (1.1) | -0.1 (1.3)
  Whole Grains (0-10 score possible, higher indicating healthier score) | 0.4 (1.8) | 0.6 (1.3)
  Dairy (0-10 score possible, higher indicating healthier score) | -0.9 (2.3) | -1.1 (2.0)
  Total Protein Foods (0-5 score possible, higher indicating healthier score) | 0.3 (0.5) | 0.0 (0.3)
  Seafood and Plant Proteins (0-5 score possible, higher indicating healthier score) | 0.6 (0.9) | 0.3 (0.9)
  Fatty Acids (0-10 score possible, higher indicating healthier score) | 0.1 (2.5) | 0.4 (2.3)
  Refined Grains (0-10 score possible, higher indicating healthier score) | -0.3 (2.4) | -2.0 (2.0)
  Sodium (0-10 score possible, higher indicating healthier score) | -1.9 (2.5) | -1.5 (2.5)
  Added Sugars (0-10 score possible, higher indicating healthier score) | 0.8 (2.0) | 0.5 (1.9)
  Saturated Fats (0-10 score possible, higher indicating healthier score) | 0.8 (2.8) | 0.7 (2.4)
  Total HEI (0-100 score possible, higher indicating healthier) | 0.3 (9.2) | -3.5 (7.9)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for an average of 12-13 weeks for all participants. This time frame is equivalent to the study length from the first/baseline visit.
Arm/Group | Lentil | Control
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 0/20 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-10-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT04283448/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/48/NCT04283448/ICF_001.pdf